CLINICAL TRIAL: NCT05861414
Title: Intervention Effect of Emotional Working Memory Training on University Students With Depressive Symptom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yu-hua Weng (Other)
Responsible Party: Sponsor-Investigator, Yu-hua Weng, Master, Fujian Medical University
Organization: Fujian Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022159
Record Dates: First submitted 2023-04-26; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Depressive Symptoms
Keywords: Emotional working memory training; Depressive symptoms
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 21 days of emotional working memory training
  Interventions: Behavioral: EWM-T
- control group (No Intervention)

INTERVENTIONS:
Behavioral: EWM-T — This paradigm was adapted from the n-back program described by Jaeggi et al. (2009) and comprised an affective dual n-back task consisting of a series of trials, each of which simultaneously presented a face (for 500 ms) on a 4 × 4 grid on a monitor. Intermediate interval 2500ms, during which, Participants press a button to determine if the current face or position is consistent with the first n. If the position is the same, press "F"; if the face is the same, press "J"; if the face and position are not the same, do not react.
  The faces used in this training were selected from the Chinese Facial Emotional Picture System (CFAPS), and 12 faces (six male and six female) with fear, anger, disgust, and sadness were selected as n-back experimental materials.
  Arms: Experimental group

SUMMARY:
Objective: To investigate the effects of emotional working memory training (EWM-T) on depressive symptoms and rumination among university students.

Methods: The experimental group comprised 25 participants who underwent 21 days of emotional working memory training, which involved viewing a continuous stream of negative emotional face content on a grid and remembering the faces and locations presented on the grid. The control group consisted of 25 participants. The Beck Depression Inventory-II (BDI-II), the Chinese version of the Character-Digital Breadth Test, and the Ruminative Responses Scale (RRS) were used as the pre- and post-test indicators.

DETAILED DESCRIPTION:
1. Participants and Design The G*Power 3.1 program was used to determine the recommended sample size is 46 for the study(d=0.35,1-β＝80％,α=0.05). This anticipated effect size was based on a working memory training intervention experiment, which had a medium effect size (Unread and Koster 2014).

   The participants were recruited from Fujian Medical University, and 278 students volunteered to take part in the BDI-Ⅱ. Finally, 50 university students with BDI-II scores above 14 points and with no suicidal behavior were recruited as participants. They were randomly assigned to either an experimental group (n=25) or a control group (n=25). After grouping, the participants' rumination tendency and working memory ability were assessed using the Ruminative Responses Scale (RRS) and the Character-Digital Breadth Test.

   Subsequently, the experimental group completed twenty-one 20 to 30 minute EWM-T training sessions within one month, and the control group was not treated. A month later, the participants were assessed again for depressive symptoms, working memory ability, and rumination tendency.

   This study was approved by the Ethics Committee of Fujian Medical University, and all the participants provided signed informed consent. If they were found to be at risk of suicide, the experiment was terminated immediately. If the participants felt uncomfortable, they could withdraw from the experiment at any time, and psychological help was provided if they so desired.
2. Materials and Measures 2.1 Beck Depression Inventory-Ⅱ (BDI-Ⅱ) The BDI-II is the most prevalent self-report scale assessing the presence and severity of depressive symptoms. It is a 21-item scale that was used to assess the severity of depressive symptoms in the past two weeks. The scores range from 0 to 63. A higher total score on the scale indicated more severe depressive symptoms. (Wang 2011).

   2.2 Ruminative Responses Scale (RRS) The Ruminative Response Scale (RRS) is a scale of 22 items scored on a 4-point Likert scale ranging from 1 (almost never) to 4 (almost always). It was used to assess ruminative thinking, with higher scores indicating a higher degree of ruminative symptoms. It includes three dimensions: symptom rumination, forced thinking, and introspective. The Chinese version of the RRS is suitable for evaluating the rumination thinking of Chinese university students (Han and Yang 2009).

   2.3 Character-Digital Breadth Test The experimenter read aloud some combinations of characters and numbers, and after the experimenter finished speaking, the participants first stated the numbers in descending order and then the characters in descending order. For example, in the fourth pass: "8B3A," the participant needed to answer "38AB," and then the test began after the person understood the rules. Different levels (2-9 levels) had various lengths of characters and numbers. The higher the level, the longer the length. Each level contained four items. Scoring was based on the total number of correct items passed (correct number of character digit spans) and the rank of the longest items passed (longest sequence of character digit spans). Each item was completed when all items at a certain level were incorrect. The greater the number of correct items passed, the higher the level of the longest items, the greater the working memory breadth, and the stronger the working memory ability .

   2.4 EWM-T This paradigm was adapted from the n-back program described by Jaeggi et al. (2009) and comprised an affective dual n-back task consisting of a series of trials, each of which simultaneously presented a face (for 500 ms) on a 4 × 4 grid on a monitor. Intermediate interval 2500ms, during which, Participants press a button to determine if the current face or position is consistent with the first n. If the position is the same, press "F"; if the face is the same, press "J"; if the face and position are not the same, do not react.

   Training started at n = 1; if the participants got more than 80% correct, the level of n-back increased by one in the next block. Conversely, if the participants got less than 60% correct, the level of n-back decreased by 1 in the next block. If the 2-back accuracy was greater than 80%, the next block difficulty was upgraded to 3-back; if the 3-back accuracy was less than 60%, the next block difficulty was downgraded to 2-back. The maximum value of n is 8. The 20 daily 20-30 min training sessions consisted of 20 blocks of 20+ n trials.

   The faces used in this training were selected from the Chinese Facial Emotional Picture System (CFAPS), and 12 faces (six male and six female) with fear, anger, disgust, and sadness were selected as n-back experimental materials.
3. Data Analysis An independent samples t-test was used to determine whether the experimental and control groups had varying levels of BDI-II, RRS, and Character-Digital Breadth Test scores at baseline and post-test. T-test determined whether there were significant changes in BDI-II, RRS, and Character-Digital Breadth Test scores from pre-test to post-test in the experimental and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Study from Fujian Medical University, BDI-II scores above 14 points.

Exclusion Criteria:

* no suicidal behavior

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory-II (BDI-II) score | one month
  Beck Depression Inventory-Ⅱ is the most prevalent self-report scale assessing the presence and severity of depressive symptoms. It is a 21-item scale that was used to assess the severity of depressive symptoms in the past two weeks. The scores range from 0 to 63. A higher total score on the scale indicated more severe depressive symptoms.
Ruminative Responses Scale (RRS) score | one month
  The Ruminative Response Scale (RRS) is a scale of 22 items scored on a 4-point Likert scale ranging from 1 (almost never) to 4 (almost always). It was used to assess ruminative thinking, with higher scores indicating a higher degree of ruminative symptoms. It includes three dimensions: symptom rumination, forced thinking, and introspective.
The Chinese version of the Character-Digital Breadth Test score | one month
  The experimenter read aloud some combinations of characters and numbers, and after the experimenter finished speaking, the participants first stated the numbers in descending order and then the characters in descending order. For example, in the fourth pass: "8B3A," the participant needed to answer "38AB," and then the test began after the person understood the rules. Different levels (2-9 levels) had various lengths of characters and numbers. The higher the level, the longer the length. Each level contained four items. Scoring was based on the total number of correct items passed (correct number of character digit spans) and the rank of the longest items passed (longest sequence of character digit spans). Each item was completed when all items at a certain level were incorrect. The greater the number of correct items passed, the higher the level of the longest items, the greater the working memory breadth, and the stronger the working memory ability .

CONTACTS AND LOCATIONS:
Locations (1):
- School of Health, Fujian Medical University, Fuzhou, China

IPD SHARING:
Plan to Share IPD: Undecided
Do not understand Share IPD